CLINICAL TRIAL: NCT06324188
Title: Early Atrial Fibrillation Ablation for Stroke Prevention in Patients With High Comorbidity Burden (EASThigh-AFNET 11)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EASThigh-AFNET 11
Record Dates: First submitted 2024-03-04; First posted 2024-03-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
Keywords: Early atrial fibrillation ablation; High comorbidity burden; CHA2DS2-VASc score; Early rhythm control; Stroke; Heart failure; Cardiovascular death; Cryoballoon
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: blinded endpoint assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early atrial fibrillation ablation (Other)
  Interventions: Other: Early atrial fibrillation ablation
- Usual Care (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Early atrial fibrillation ablation — Patients randomised to early atrial fibrillation ablation will undergo pulmonary vein isolation within 2 months after randomisation.
  Arms: Early atrial fibrillation ablation
Other: Usual Care — Usual care will consist of optimal AF therapy based on guideline recommendations and local protocols and usage.The choice of therapies and medications follows routine care in line with medical guidelines and local policies at the discretion of the treating physician and should be based on the individual medical status of each study patient.
  Arms: Usual Care

SUMMARY:
EASThigh-AFNET 11 is an international, prospective, randomized, open, blinded endpoint assessment, multicenter trial (Treatment Strategy trial).

The objective of EASThigh-AFNET 11 is to investigate whether early atrial fibrillation ablation in patients with atrial fibrillation (AF) and a high comorbidity burden (CHA2DS2-VASc ≥4) reduces cardiovascular events (stroke, cardiovascular death, or heart failure events) compared to usual care.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is associated with high morbidity and mortality. Even on optimal anticoagulation and therapy of concomitant conditions, many patients with AF suffer cardiovascular events, especially heart failure events, stroke, and cardiovascular death. Most of these events occur in elderly patients with comorbidities. Early rhythm control, mainly delivered using antiarrhythmic drugs, reduces AF-related complications when added to anticoagulation, rate control, and treatment of comorbidities when compared to current practice that offers rhythm control mainly to reduce symptoms. The outcome-reducing effect of early rhythm control is most pronounced in patients with multiple comorbidities, quantified by a CHA2DS2-VASc score ≥ 4. Attaining sinus rhythm is the key mediator for the outcome-reducing effect of early rhythm control. Atrial fibrillation ablation controls the rhythm better than drug-based rhythm control, avoids long-term antiarrhythmic drug treatment, thus reducing polypharmacy, and may therefore be the ideal rhythm control treatment in patients with AF and a high comorbidity burden. This hypothesis needs testing. The investigator-initiated EASThigh-AFNET 11 trial evaluates the effectiveness and safety of early atrial fibrillation ablation in patients with recently diagnosed AF and a high comorbidity burden.

EASThigh-AFNET 11 is a Treatment Strategy trial randomizing 2312 patients with AF and a high comorbidity burden to early atrial fibrillation ablation or usual care to achieve a fixed number of primary endpoint events of n=527. All therapies are clinically approved. The primary outcome is a composite of cardiovascular death, stroke, and hospitalization for worsening of heart failure. The primary safety outcome is a composite of all-cause death and serious complications of AF therapy. Secondary outcome parameters address safety, patient reported outcomes and cognitive function.

EASThigh-AFNET 11 was recommended for funding by the Expert Advisory Panel of the Global Cardiovascular Research Funders Forum (GCRFF).

ELIGIBILITY:
Inclusion Criteria:

I1. AF first diagnosed within 5 years prior to enrolment and documented in body surface ECG

I2. High comorbidity estimated by CHA2DS2-VASc score of 4 or more

I3. Patient suitable for ablation using cryoballoon ablation systems or other ablation systems with comparable efficacy and safety from Medtronic

I4. Age ≥ 18 years

I5. Provision of signed informed consent

Exclusion Criteria:

General exclusion criteria

E1. Any disease that limits life expectancy to less than 1 year.

E2. Participation in another clinical trial, either within the 3 months prior to enrolment or still on-going (participation in potential sub-studies connected to this trial is permitted).

E3. Previous participation in EASThigh-AFNET 11.

E4. Pregnant women.

E5. Breastfeeding women.

E6. Drug abuse or clinically manifest alcohol abuse.

Exclusion criteria related to a cardiac condition

E7. Prior AF ablation or surgical therapy of AF.

E8. Patients not suitable for AF ablation.

E9. Patients with a history of stroke which occurred within 3 months prior to enrolment.

E10. Valve disease requiring specific therapy.

Exclusion criteria based on laboratory abnormalities

E11. Clinically manifested thyroid dysfunction requiring therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2312 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular complications related to AF | Throughout study completion, estimated at a mean of 4 years
  It is defined as time from randomisation to the first occurrence of a composite of cardiovascular death, stroke (either ischemic or hemorrhagic), or hospitalisation for worsening of heart failure.
The primary safety outcome is a composite of all-cause death and serious complications of AF therapy. | Throughout study completion, estimated at a mean of 4 years
  Serious Adverse Events (SAEs), including primary and secondary outcome parameters if based on clinical events, will be adjudicated by the independent Clinical Event Committee (CEC) according to standardised definitions given in the CEC charter.

SECONDARY OUTCOMES:
Number of nights spent in hospital | Throughout study completion, estimated at a mean of 4 years
Time from randomisation to first occurrence of each of the individual components of the primary outcome | Throughout study completion, estimated at a mean of 4 years
All-cause death | Throughout study completion, estimated at a mean of 4 years
Serious adverse events related to AF therapy | Throughout study completion, estimated at a mean of 4 years
Time from randomisation to first cardiovascular hospitalisation | Throughout study completion, estimated at a mean of 4 years
Number of cardiovascular hospitalisations (over-night stay) | Throughout study completion, estimated at a mean of 4 years
Changes in left ventricular ejection fraction | comparing baseline with 24 months follow up (FU)
Changes in quality of life | comparing baseline with 12 and 24 months FU
  assessed by EQ-5D-5L
Changes in quality of life | comparing baseline with 12 and 24 months FU
  assessed by AFEQT
Changes in cognitive function | comparing baseline with 24 months FU
  assessed by Montreal-Cognitive-Assessment-Test
Cardiac rhythm status | at 12 and 24 months FU
  sinus rhythm compared to AF
AF pattern | at 12 and 24 months FU
Time from randomisation to first clinical recurrence of AF | Throughout study completion, estimated at a mean of 4 years
Time from randomisation to first progression of AF | Throughout study completion, estimated at a mean of 4 years
  i. e. from paroxysmal to persistent or longstanding persistent or permanent and each of these components

CONTACTS AND LOCATIONS:
Overall Officials: Paulus Kirchhof, Prof. Dr., Study Director — University Heart and Vascular Center Hamburg, University Hospital Hamburg Eppendorf; Andreas Rillig, PD Dr., Study Director — University Heart and Vascular Center Hamburg, University Hospital Hamburg Eppendorf; Jason Andrade, Prof. Dr., Principal Investigator — University of British Columbia, Vancouver General Hospital, Department of Electrophysiology; André Ng, Prof. Dr., Principal Investigator — Department of Cardiovascular Sciences, University of Leicester; Prash Sanders, Prof. Dr., Principal Investigator — Centre for Heart Rhythm Disorders, University of Adelaide, Royal Adelaide Hospital; Volker Straub, Principal Investigator — Patient representative; Kevin Vernooy, Prof. Dr., Principal Investigator — Department of Cardiology, Cardiovascular Research Institute Maastricht (CARIM), Maastricht University Medical Center (MUMC); Antonia Zapf, Prof. Dr., Principal Investigator — Institute of Medical Biometry and Epidemiology, University Medical Center Hamburg-Eppendorf
Locations (7):
- Several sites, Multiple Locations, Australia
- Several sites, Multiple Locations, Canada
- Several sites, Multiple Locations, Germany
- Several sites, Multiple Locations, Netherlands
- Several sites, Multiple Locations, Poland
- Several sites, Multiple Locations, Spain
- Several sites, Multiple Locations, United Kingdom

REFERENCES:
- [Background] Kirchhof P, Camm AJ, Goette A, Brandes A, Eckardt L, Elvan A, Fetsch T, van Gelder IC, Haase D, Haegeli LM, Hamann F, Heidbuchel H, Hindricks G, Kautzner J, Kuck KH, Mont L, Ng GA, Rekosz J, Schoen N, Schotten U, Suling A, Taggeselle J, Themistoclakis S, Vettorazzi E, Vardas P, Wegscheider K, Willems S, Crijns HJGM, Breithardt G; EAST-AFNET 4 Trial Investigators. Early Rhythm-Control Therapy in Patients with Atrial Fibrillation. N Engl J Med. 2020 Oct 1;383(14):1305-1316. doi: 10.1056/NEJMoa2019422. Epub 2020 Aug 29. PMID 32865375
- [Background] Rillig A, Borof K, Breithardt G, Camm AJ, Crijns HJGM, Goette A, Kuck KH, Metzner A, Vardas P, Vettorazzi E, Wegscheider K, Zapf A, Kirchhof P. Early Rhythm Control in Patients With Atrial Fibrillation and High Comorbidity Burden. Circulation. 2022 Sep 13;146(11):836-847. doi: 10.1161/CIRCULATIONAHA.122.060274. Epub 2022 Aug 15. PMID 35968706
- [Background] Eckardt L, Sehner S, Suling A, Borof K, Breithardt G, Crijns H, Goette A, Wegscheider K, Zapf A, Camm J, Metzner A, Kirchhof P. Attaining sinus rhythm mediates improved outcome with early rhythm control therapy of atrial fibrillation: the EAST-AFNET 4 trial. Eur Heart J. 2022 Oct 21;43(40):4127-4144. doi: 10.1093/eurheartj/ehac471. PMID 36036648
- [Background] Andrade JG, Wells GA, Deyell MW, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Macle L, Verma A; EARLY-AF Investigators. Cryoablation or Drug Therapy for Initial Treatment of Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):305-315. doi: 10.1056/NEJMoa2029980. Epub 2020 Nov 16. PMID 33197159
- [Background] Andrade JG, Deyell MW, Macle L, Wells GA, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Cadrin-Tourigny J, Kochhauser S, Verma A; EARLY-AF Investigators. Progression of Atrial Fibrillation after Cryoablation or Drug Therapy. N Engl J Med. 2023 Jan 12;388(2):105-116. doi: 10.1056/NEJMoa2212540. Epub 2022 Nov 7. PMID 36342178
- [Background] Dickow J, Kirchhof P, Van Houten HK, Sangaralingham LR, Dinshaw LHW, Friedman PA, Packer DL, Noseworthy PA, Yao X. Generalizability of the EAST-AFNET 4 Trial: Assessing Outcomes of Early Rhythm-Control Therapy in Patients With Atrial Fibrillation. J Am Heart Assoc. 2022 Jun 7;11(11):e024214. doi: 10.1161/JAHA.121.024214. Epub 2022 May 27. PMID 35621202
- [Background] Dickow J, Kany S, Roth Cardoso V, Ellinor PT, Gkoutos GV, Van Houten HK, Kirchhof P, Metzner A, Noseworthy PA, Yao X, Rillig A. Outcomes of Early Rhythm Control Therapy in Patients With Atrial Fibrillation and a High Comorbidity Burden in Large Real-World Cohorts. Circ Arrhythm Electrophysiol. 2023 May;16(5):e011585. doi: 10.1161/CIRCEP.122.011585. Epub 2023 Mar 21. PMID 36942567